CLINICAL TRIAL: NCT02846389
Title: Randomized Controlled Trial of Exercise to Reduce Cancer Related Fatigue in Women Undergoing Radiation Treatment for Breast Cancer
Brief Title: Trial of Exercise to Reduce Cancer Related Fatigue in Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Lombardi Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2016-0162
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cancer Related Fatigue
Keywords: Radiation therapy for Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Exercise (Experimental): Moderate exercise - 15 minutes a day using a pedal box before or after radiation at the hospital (75 minutes a week).
  Interventions: Other: Moderate Exercise
- Control Group (No Intervention): No exercise

INTERVENTIONS:
Other: Moderate Exercise — Aerobic training utilizing the portable stationary pedal exerciser (Pedlar) which contains two cycling pedals mounted to a stationary block that allows patients to exercise while sitting. Participants are required to perform 15 minutes/day of aerobic exercise using the Pedlar device on radiation treatment days; during a standard radiation course, this will typically yield 75 minutes/week of aerobic time.
  Arms: Moderate Exercise

SUMMARY:
Like other cancer treatments, radiation therapy can make people feel fatigued, or tired. The investigators think that moderate exercise, done 15 minutes at a time, can reduce the fatigue. This study is designed to gather more information, so that in the future, doctors can recommend whether patients should engage in exercise during a radiation treatment course.

DETAILED DESCRIPTION:
Cancer related fatigue (CRF) is a common and debilitating side effect of radiotherapy in breast cancer patients. Physical activity interventions can attenuate CRF. The proposed study is a randomized, controlled trial (RCT) of exercise of structured moderate-intensity exercise intervention, delivered concurrently with radiotherapy, to reduce CRF and improve health-related quality of life among breast cancer patients. Eighty women with breast cancer scheduled to receive radiation therapy at Hackensack University Medical Center (HUMC) will be randomized to one of the two trial arms:1) a facility-based aerobic exercise utilizing a portable stationary pedal exerciser; or 2) a control group. Intervention arm participants will exercise at the hospital either before or after their radiation treatment. Assessments will be conducted at baseline, 4 weeks into radiation course, and at 4-week follow-up visit. The outcome variables are CRF, biomarkers of inflammation, and health-related quality of life (QOL). The study will provide preliminary evidence on whether a short-term moderate-intensity exercise intervention might be effective in reducing CRF in women undergoing radiotherapy for breast cancer, and whether this effect is mediated by inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. women between the ages of 18 and 75 years
2. histologically confirmed non-metastatic carcinoma of the breast (in situ disease or invasive)
3. radiation therapy naïve
4. sedentary activity level at baseline, as defined by less than 60 minutes per week of modest physical activity based on 7-day physical activity recall questionnaire
5. ambulatory
6. negative serum pregnancy test and not planning to become pregnant in the next three months
7. able to provide meaningful consent.
8. Patients must have been deemed by their medical oncologist or internist that they "may participate in [this] exercise trial." Prior to randomization, participants are required to complete a Physical Activity Readiness Questionnaire (PAR-Q) that includes questions regarding physical and medical conditions that would preclude safe participation in an exercise program.

Exclusion Criteria:

1. younger than 18 or older than 75 years
2. no histological confirmation of breast cancer
3. prior breast, chest, or pelvic radiotherapy
4. concurrent chemotherapy
5. distant metastases
6. physical limitations that contraindicate participation in low to moderate intensity exercise
7. positive pregnancy test
8. currently engaged in moderate to vigorous physical activity
9. psychiatric disorder which would render the participant unable to provide informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2017-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Lewis, M.D., Ph.D, Principal Investigator — Hackensack UMC
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Potthoff K, Schmidt ME, Wiskemann J, Hof H, Klassen O, Habermann N, Beckhove P, Debus J, Ulrich CM, Steindorf K. Randomized controlled trial to evaluate the effects of progressive resistance training compared to progressive muscle relaxation in breast cancer patients undergoing adjuvant radiotherapy: the BEST study. BMC Cancer. 2013 Mar 28;13:162. doi: 10.1186/1471-2407-13-162. PMID 23537231
- [Background] Fisher B, Jeong JH, Anderson S, Bryant J, Fisher ER, Wolmark N. Twenty-five-year follow-up of a randomized trial comparing radical mastectomy, total mastectomy, and total mastectomy followed by irradiation. N Engl J Med. 2002 Aug 22;347(8):567-75. doi: 10.1056/NEJMoa020128. PMID 12192016
- [Background] Zelefsky MJ, Fuks Z, Hunt M, Yamada Y, Marion C, Ling CC, Amols H, Venkatraman ES, Leibel SA. High-dose intensity modulated radiation therapy for prostate cancer: early toxicity and biochemical outcome in 772 patients. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1111-6. doi: 10.1016/s0360-3016(02)02857-2. PMID 12128109
- [Background] Fisher B, Dignam J, Wolmark N, Mamounas E, Costantino J, Poller W, Fisher ER, Wickerham DL, Deutsch M, Margolese R, Dimitrov N, Kavanah M. Lumpectomy and radiation therapy for the treatment of intraductal breast cancer: findings from National Surgical Adjuvant Breast and Bowel Project B-17. J Clin Oncol. 1998 Feb;16(2):441-52. doi: 10.1200/JCO.1998.16.2.441. PMID 9469327
- [Background] Bagshaw MA, Kaplan ID, Cox RC. Prostate cancer. Radiation therapy for localized disease. Cancer. 1993 Feb 1;71(3 Suppl):939-52. doi: 10.1002/1097-0142(19930201)71:3+3.0.co;2-0. PMID 8428344
- [Background] Alcantara-Silva TR, Freitas-Junior R, Freitas NM, Machado GD. Fatigue related to radiotherapy for breast and/or gynaecological cancer: a systematic review. J Clin Nurs. 2013 Oct;22(19-20):2679-86. doi: 10.1111/jocn.12236. Epub 2013 May 8. PMID 23651041
- [Background] Steindorf K, Schmidt ME, Klassen O, Ulrich CM, Oelmann J, Habermann N, Beckhove P, Owen R, Debus J, Wiskemann J, Potthoff K. Randomized, controlled trial of resistance training in breast cancer patients receiving adjuvant radiotherapy: results on cancer-related fatigue and quality of life. Ann Oncol. 2014 Nov;25(11):2237-2243. doi: 10.1093/annonc/mdu374. Epub 2014 Aug 5. PMID 25096607
- [Background] Dhruva A, Dodd M, Paul SM, Cooper BA, Lee K, West C, Aouizerat BE, Swift PS, Wara W, Miaskowski C. Trajectories of fatigue in patients with breast cancer before, during, and after radiation therapy. Cancer Nurs. 2010 May-Jun;33(3):201-12. doi: 10.1097/NCC.0b013e3181c75f2a. PMID 20357659
- [Background] Jereczek-Fossa BA, Marsiglia HR, Orecchia R. Radiotherapy-related fatigue. Crit Rev Oncol Hematol. 2002 Mar;41(3):317-25. doi: 10.1016/s1040-8428(01)00143-3. PMID 11880207
- [Background] Morrow GR, Shelke AR, Roscoe JA, Hickok JT, Mustian K. Management of cancer-related fatigue. Cancer Invest. 2005;23(3):229-39. doi: 10.1081/cnv-200055960. PMID 15945509
- [Background] Mustian KM, Peppone L, Darling TV, Palesh O, Heckler CE, Morrow GR. A 4-week home-based aerobic and resistance exercise program during radiation therapy: a pilot randomized clinical trial. J Support Oncol. 2009 Sep-Oct;7(5):158-67. PMID 19831159
- [Background] Noal S, Levy C, Hardouin A, Rieux C, Heutte N, Segura C, Collet F, Allouache D, Switsers O, Delcambre C, Delozier T, Henry-Amar M, Joly F. One-year longitudinal study of fatigue, cognitive functions, and quality of life after adjuvant radiotherapy for breast cancer. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):795-803. doi: 10.1016/j.ijrobp.2010.06.037. Epub 2010 Oct 1. PMID 20888704
- [Background] Hickok JT, Roscoe JA, Morrow GR, Mustian K, Okunieff P, Bole CW. Frequency, severity, clinical course, and correlates of fatigue in 372 patients during 5 weeks of radiotherapy for cancer. Cancer. 2005 Oct 15;104(8):1772-8. doi: 10.1002/cncr.21364. PMID 16116608
- [Background] Ryan JL, Carroll JK, Ryan EP, Mustian KM, Fiscella K, Morrow GR. Mechanisms of cancer-related fatigue. Oncologist. 2007;12 Suppl 1:22-34. doi: 10.1634/theoncologist.12-S1-22. PMID 17573453
- [Background] Bower JE, Ganz PA, Tao ML, Hu W, Belin TR, Sepah S, Cole S, Aziz N. Inflammatory biomarkers and fatigue during radiation therapy for breast and prostate cancer. Clin Cancer Res. 2009 Sep 1;15(17):5534-40. doi: 10.1158/1078-0432.CCR-08-2584. Epub 2009 Aug 25. PMID 19706826
- [Background] Geinitz H, Zimmermann FB, Stoll P, Thamm R, Kaffenberger W, Ansorg K, Keller M, Busch R, van Beuningen D, Molls M. Fatigue, serum cytokine levels, and blood cell counts during radiotherapy of patients with breast cancer. Int J Radiat Oncol Biol Phys. 2001 Nov 1;51(3):691-8. doi: 10.1016/s0360-3016(01)01657-1. PMID 11597810
- [Background] Lundh Hagelin C, Wengstrom Y, Furst CJ. Patterns of fatigue related to advanced disease and radiotherapy in patients with cancer-a comparative cross-sectional study of fatigue intensity and characteristics. Support Care Cancer. 2009 May;17(5):519-26. doi: 10.1007/s00520-008-0502-5. Epub 2008 Sep 13. PMID 18791747
- [Background] Hovdenak N, Fajardo LF, Hauer-Jensen M. Acute radiation proctitis: a sequential clinicopathologic study during pelvic radiotherapy. Int J Radiat Oncol Biol Phys. 2000 Nov 1;48(4):1111-7. doi: 10.1016/s0360-3016(00)00744-6. PMID 11072170
- [Background] Larsen A, Bjorge B, Klementsen B, Helgeland L, Wentzel-Larsen T, Fagerhol MK, Hovdenak N, Dahl O. Time patterns of changes in biomarkers, symptoms and histopathology during pelvic radiotherapy. Acta Oncol. 2007;46(5):639-50. doi: 10.1080/02841860601099241. PMID 17562440
- [Background] Symon Z, Goldshmidt Y, Picard O, Yavzori M, Ben-Horin S, Alezra D, Barshack I, Chowers Y. A murine model for the study of molecular pathogenesis of radiation proctitis. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):242-50. doi: 10.1016/j.ijrobp.2009.07.1736. PMID 20005457
- [Background] Greenberg DB, Gray JL, Mannix CM, Eisenthal S, Carey M. Treatment-related fatigue and serum interleukin-1 levels in patients during external beam irradiation for prostate cancer. J Pain Symptom Manage. 1993 May;8(4):196-200. doi: 10.1016/0885-3924(93)90127-h. PMID 7963760
- [Background] Christiansen H, Saile B, Hermann RM, Rave-Frank M, Hille A, Schmidberger H, Hess CF, Ramadori G. Increase of hepcidin plasma and urine levels is associated with acute proctitis and changes in hemoglobin levels in primary radiotherapy for prostate cancer. J Cancer Res Clin Oncol. 2007 May;133(5):297-304. doi: 10.1007/s00432-006-0170-0. Epub 2006 Nov 25. PMID 17393200
- [Background] Saligan LN, Kim HS. A systematic review of the association between immunogenomic markers and cancer-related fatigue. Brain Behav Immun. 2012 Aug;26(6):830-48. doi: 10.1016/j.bbi.2012.05.004. Epub 2012 May 14. PMID 22595751
- [Background] Courneya KS, Mackey JR, Bell GJ, Jones LW, Field CJ, Fairey AS. Randomized controlled trial of exercise training in postmenopausal breast cancer survivors: cardiopulmonary and quality of life outcomes. J Clin Oncol. 2003 May 1;21(9):1660-8. doi: 10.1200/JCO.2003.04.093. PMID 12721239
- [Background] Cuesta-Vargas AI, Buchan J, Arroyo-Morales M. A multimodal physiotherapy programme plus deep water running for improving cancer-related fatigue and quality of life in breast cancer survivors. Eur J Cancer Care (Engl). 2014 Jan;23(1):15-21. doi: 10.1111/ecc.12114. Epub 2013 Aug 16. PMID 23947581
- [Background] Galanti G, Stefani L, Gensini G. Exercise as a prescription therapy for breast and colon cancer survivors. Int J Gen Med. 2013 Apr 16;6:245-51. doi: 10.2147/IJGM.S42720. Print 2013. PMID 23620675
- [Background] Blanchard CM, Courneya KS, Laing D. Effects of acute exercise on state anxiety in breast cancer survivors. Oncol Nurs Forum. 2001 Nov-Dec;28(10):1617-21. PMID 11759309
- [Background] Byrne A, Byrne DG. The effect of exercise on depression, anxiety and other mood states: a review. J Psychosom Res. 1993 Sep;37(6):565-74. doi: 10.1016/0022-3999(93)90050-p. PMID 8410742
- [Background] King AC, Taylor CB, Haskell WL. Effects of differing intensities and formats of 12 months of exercise training on psychological outcomes in older adults. Health Psychol. 1993 Jul;12(4):292-300. doi: 10.1037//0278-6133.12.4.292. PMID 8404803
- [Background] Blumenthal JA, Williams RS, Needels TL, Wallace AG. Psychological changes accompany aerobic exercise in healthy middle-aged adults. Psychosom Med. 1982 Dec;44(6):529-36. doi: 10.1097/00006842-198212000-00004. PMID 7163456
- [Background] Singh NA, Clements KM, Fiatarone MA. A randomized controlled trial of progressive resistance training in depressed elders. J Gerontol A Biol Sci Med Sci. 1997 Jan;52(1):M27-35. doi: 10.1093/gerona/52a.1.m27. PMID 9008666
- [Background] MacVicar MG, Winningham ML, Nickel JL. Effects of aerobic interval training on cancer patients' functional capacity. Nurs Res. 1989 Nov-Dec;38(6):348-51. PMID 2587289
- [Background] Mock V, Frangakis C, Davidson NE, Ropka ME, Pickett M, Poniatowski B, Stewart KJ, Cameron L, Zawacki K, Podewils LJ, Cohen G, McCorkle R. Exercise manages fatigue during breast cancer treatment: a randomized controlled trial. Psychooncology. 2005 Jun;14(6):464-77. doi: 10.1002/pon.863. PMID 15484202
- [Background] Monga U, Garber SL, Thornby J, Vallbona C, Kerrigan AJ, Monga TN, Zimmermann KP. Exercise prevents fatigue and improves quality of life in prostate cancer patients undergoing radiotherapy. Arch Phys Med Rehabil. 2007 Nov;88(11):1416-22. doi: 10.1016/j.apmr.2007.08.110. PMID 17964881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Exercise | Control Group
Started | 11 | 13
Completed | 10 | 12
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Exercise | Control Group | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 1 | 3 | 4
Age, Continuous [Median (Full Range); unit: years] | 54 [38 to 72] | 51 [40 to 65] | 53.5 [38 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Change in Fatigue Via Functional Assessment of Chronic Illness Therapy (FACIT-Fatigue) Survey Instrument.
Description: The Functional Assessment of Chronic Illness Therapy (FACIT) is a 13-item subscale developed to identify a finite set of concerns specific to fatigue. The responses to the 13 items on the FACIT-Fatigue questionnaire are each measured on a 4-point likert scale, with score ranging from 0 to 52 (52 being the total score allowed). The FACIT-Fatigue scale has been validated in patients with cancer and showed excellent internal consistency and reliability.
  Responses to questions are scored: Not at all (0), A little bit (1), Somewhat (2) Quite a bit (3), Very much (4). Some scores are reversed depending on the question. The sum of the item scores are multiplied by the number of items in the scale, then divide by the number of items answered. This produces the score. The higher the score, the better the QOL.
Time Frame: Baseline, 4 weeks into RT
Measure: Mean (Standard Deviation); unit: FACIT Score
Arm/Group | Moderate Exercise | Control Group
Number analyzed (Participants) | 11 | 13
FACIT Score
  Baseline | 17 (11) | 14 (8)
  4 weeks into RT | 21 (9) | 18 (14)

2. Primary Outcome: Assessment of Change in Blood Biomarker of Inflammation: High Sensitivity CRP (hsCRP)
Description: Serum hsCRP will be measured on the Vitros 5,1 FS Chemistry platform via an immunoassay with a reportable range of 0.10 -15.00 mg/L, and intra- and inter-assay CVs of 1.8-4.0%. Change is reported based on the difference in the group mean of Serum hsCRP level between baseline and T4 visit.
Time Frame: Baseline, 4 weeks into RT
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Moderate Exercise | Control Group
Number analyzed (Participants) | 11 | 13
milligrams per liter (mg/L)
  Baseline | 0.39 (0.47) | 0.29 (0.33)
  4 weeks into RT | 0.21 (0.19) | 0.13 (0.14)

3. Primary Outcome: Assessment of Change in Blood Biomarker of Inflammation: Serum Fibrinogen
Description: Fibrinogen will be measured using standardized clinical protocols. All assays have intra- and inter-assays coefficient of variations <10%. Change is reported based on the difference in the group mean of Serum fibrinogen level between baseline and T4 visit.
Time Frame: Baseline, 4 weeks into RT
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Moderate Exercise | Control Group
Number analyzed (Participants) | 11 | 13
milligrams per deciliter (mg/dL)
  Baseline | 326 (69) | 307 (116)
  4 weeks into RT | 288 (78) | 296 (77)

4. Primary Outcome: Assessment of Change in Blood Biomarker of Inflammation: Ferritin
Description: Ferritin will be measured using standardized clinical protocols. All assays have intra- and inter-assays coefficient of variations <10%. Change is reported based on the difference in the group mean of ferritin levels between baseline and T4 visit.
Time Frame: Baseline, 4 weeks into RT
Measure: Mean (Standard Deviation); unit: Micrograms per liter (mcg/L)
Arm/Group | Moderate Exercise | Control Group
Number analyzed (Participants) | 11 | 13
Micrograms per liter (mcg/L)
  Baseline | 0.009 (0.005) | 0.005 (0.006)
  4 weeks into RT | 0.008 (0.003) | 0.006 (0.004)

5. Secondary Outcome: Assessment of Change in Cancer-related Healthcare Quality of Life (HRQOL) Measured Using the Functional Assessment of Cancer Therapy (FACT) System Questionnaires.
Description: The Health-related quality of life (HRQOL) measures four different domains (physical well-being, functional well-being, emotional well-being, and social/family well-being). Functional Assessment of Cancer Therapy (FACT-B) is a breast cancer specific module that will be used to reflect patients' concerns; moreover, they are reliable, reproducible, and have been validated in numerous studies. Score ranging from 0 to 148 (148 being the total score allowed).
  Responses to questions are scored: Not at all (0), A little bit (1), Somewhat (2) Quite a bit (3), Very much (4). Some scores are reveresed depending on the question. The sum of the item scores are multiplied by the number of items in the scale, then divide by the number of items answered. This produces the score. The higher the score, the better the QOL.
  Change in the group sum of the FACT score between baseline and T4 visit.
Time Frame: Baseline, 4 weeks into RT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate Exercise | Control Group
Number analyzed (Participants) | 11 | 13
units on a scale
  Baseline | 70 (8) | 69 (8)
  4 weeks into RT | 66 (11) | 71 (10)

6. Other Pre Specified Outcome: Complete Blood Count Data (CBC)
Description: We will collect CBC data at each blood draw for correlative and explorative purposes.
Time Frame: Baseline, 4 weeks into RT, 4 week follow up visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Event Assessment performed through 4-week follow-up visit, an average of 14 weeks
Arm/Group | Moderate Exercise | Control Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT02846389/Prot_SAP_000.pdf